CLINICAL TRIAL: NCT04702087
Title: Randomized, Placebo-controlled Clinical Study to Evaluate the Effect of 2 Months of Nutritional Support Based on Omega 3, Leucine, Probiotic Lactobacillus Paracasei PS23 (OLEP Study) on Muscle Mass in Sarcopenic Subjects
Brief Title: Omega 3, Leucine, Probiotic Lactobacillus Paracasei PS23 on Muscle Mass in Sarcopenic Subjects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda di Servizi alla Persona di Pavia (Other)
Collaborators: Abiogen Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 202000070742
Record Dates: First submitted 2021-01-05; First posted 2021-01-08 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-09

CONDITIONS: Sarcopenia; Elderly; Omega 3
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OLEP (Experimental): Omega 3 (500 mg), leucine (2,5 g), probiotic Lactobacillus paracasei PS23
  Interventions: Dietary Supplement: OLEP
- Placebo (Placebo Comparator): isocaloric formula
  Interventions: Combination Product: Placebo

INTERVENTIONS:
Dietary Supplement: OLEP — omega 3 (500 mg), leucine (2,5 g), probiotic Lactobacillus paracasei PS23
  Arms: OLEP
Combination Product: Placebo — Isocaloric formula
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the effect of supplementation with a nutritional blend based on Omega 3 fatty acids, the probiotic leucine Lactobacillus paracasei PS23 (OLEP), on muscle mass recovery in sarcopenic patients.

ELIGIBILITY:
Inclusion Criteria:

* Sarcopenic patients (diagnosis made according to the criteria Revised European Consensus on Definition and Diagnosis)
* Body Mass Index between 20 and 30 Kg/m2

Exclusion Criteria:

* severe renal failure (glomerular filtration rate < 30 mL/min)
* moderate to severe liver failure (Child-Pugh class B or C)
* endocrine diseases associated with calcium metabolism disorders (except osteoporosis)
* known psychiatric disorders
* cancer (over the past 5 years)
* hypersensitivity to any component of the investigational nutritional supplement and
* taking to protein/amino acid supplements (up to 3 months before starting the study)
* patients unable to take oral therapy
* receiving or with indication for artificial nutrition
* who had been included in another clinical nutrition trial

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2021-01-22 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Changes on muscle mass | Baseline / 30 days / 60 days
  Evaluation of fat free mass (g)

SECONDARY OUTCOMES:
Changes on body composition | Baseline / 30 days / 60 days
  Evaluation of fat mass (g) and visceral adipose tissue (g)
Changes on physical performancy | Baseline / 60 days
  Evaluation of Tinetti scale (point scale) that measures characteristics associated with falls, assessing balance (14 items; 24 points), and gait (10 items; 16 points) for a total score up to 40 (the higher the score, the better the performance)
Changes on physical performancy | Baseline / 60 days
  Evaluation of Short Physical Performance Battery (point scale) which consists of three components: gait speed, chair-stand test, timed up and go (TUG) test (which assesses the time taken to rise from an arm chair, walk 3 m, turn, walk back, and sit down again), and balance (three different tests assessing ability to stand with the feet together in the side-by-side, semi-tandem, and tandem positions); accordingly, each component was scored from 0 (not possible) to 4 (best performance) and the scores add up to a total score ranging from 0 to 12.
Changes on functional status | Baseline / 60 days
  Evaluation of Barthel Index (point scale) (covering all the aspects of self-care independence in daily living activities, including transfer, walking, stairs, toilet use, dressing, feeding, bladder, bowel, grooming, and bathing; score range, 0 (completely dependent) -100 (complete self-sufficiency))
Changes on functional status | Baseline / 60 days
  Evaluation of activities of daily living score (point scale): a simplified scale that provides for the assignment of a point for each independent function in order to obtain a total performance result ranging from 0 (complete dependence) to 6 (independence in all functions).
Changes on muscle strength | Baseline / 30 days / 60 days
  Evaluation of muscle strength (kg)
Changes on Quality of life | Baseline / 60 days
  Evaluation of Short-Form 12-Item Health Survey (poin survey): a generic health-status measure (physical component summary score and the mental component summary score) by addressing eight health domains (physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health. Score from 0 (bad quality) to 100 (high quality).
Changes on mood | Baseline / 60 days
  Evaluation of Geriatric Depression Scale (point scale). a 30-question test with yes/no answers. 10 - 15 Points: Probable presence of depression; 6 - 9 Points: Depression possible; 0 - 5 Points: Unlikely Depression.
Changes on blood pressure | Baseline / 60 days
  Evaluation of systolic and diastolic pressure (mm/Hg)
Changes on plasma free essential amino acids | Baseline / 60 days
  Evaluation of free essential amino acids in plasma (Leucine, Isoleucine, Valine) (micromol/L)
Changes on safety parameters | Baseline / 60 days
  Evaluation of creatinine (mg/dl)
Changes on safety parameters | Baseline / 60 days
  Evaluation of alanine aminotransferase and aspartate aminotransferase (IU/L)
Changes on safety parameters | Baseline / 60 days
  Evaluation of gamma glutamyl transferase (U/L)

CONTACTS AND LOCATIONS:
Overall Officials: Mariangela Rondanelli, Principal Investigator — Fondazione Casemiro Mondino
Locations (1):
- Azienda di Servizi alla Persona, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No